CLINICAL TRIAL: NCT03203707
Title: Early Assessment and Intervention for Adolescents at Risk for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH091177-01A1
Record Dates: First submitted 2017-06-22; First posted 2017-06-29 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Bipolar Disorder; Early Intervention
Keywords: IPSRT; early intervention; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Randomized trail comparing Data-Informed Referral (DIR) for any clinical condition detected at intake assessment versus DIR + Brief Interpersonal Social Rhythm Therapy (IPSRT)
Who Masked: Outcomes Assessor
Masking Description: Participants and parents complete clinical monitoring assessments with an evaluator blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal and Social Rhythm Therapy+DIR (Experimental): IPSRT plus referral for community treatment for any psychiatric conditions identified through the psychiatric assessment at intake.
  Interventions: Behavioral: Interpersonal and Social Rhythm Therapy
- Data-Informed Referral (DIR) (No Intervention): Referral for community treatment for any psychiatric conditions identified through the psychiatric assessment at intake.

INTERVENTIONS:
Behavioral: Interpersonal and Social Rhythm Therapy — The Brief IPSRT intervention for at-risk youth includes : 1) Psychoeducation about risk for BP ; 2) Social rhythm therapy (SRT) aiming to establish and maintain stable routines to protect against onset of mood symptoms in vulnerable individuals ; and 3) Interpersonal Psychotherapy (IPT) centering on the adolescent's feelings about having a parent with BP, and linking stressful family events to mood. The intervention is delivered in 8 in-person sessions over 6 months of treatment. Parents are involved in the psychoeducation sessions, and further involvement is determined as clinically appropriate based on age and developmental status.
  Other Names: IPSRT
  Arms: Interpersonal and Social Rhythm Therapy+DIR

SUMMARY:
Bipolar disorder is a severe and chronic illness associated with significant occupational and social impairment, enormous public health costs, and high rates of suicide. The single most potent risk factor for the development of bipolar disorder is a first-degree family member with the illness; indeed, offspring of parents with bipolar disorder are a particularly high-risk group who typically display early onset and severe course of illness. Thus, early assessment and intervention for the children of parents with bipolar disorder focused on specific, measurable, and modifiable risk factors has the potential to prevent or ameliorate the progression of bipolar disorder in those at highest risk.

DETAILED DESCRIPTION:
The most potent risk factor for the development of bipolar disorder (BP) is a first-degree family member with the illness. Thus, offspring of parents with BP are a particularly high-risk group and typically experience early illness onset, severe course, and high rates of comorbid psychiatric disorders. It is well-established that poor sleep regulation is associated with the onset of depressive and manic episodes among individuals with a biological vulnerability to mood disorder. Furthermore, evidence supports sleep disturbance in at-risk youth who have not yet developed threshold mood disorders. The proposed study aims to address this core disturbance that we argue puts at-risk youth at even greater risk for development of BP-sleep and social rhythm disruption. Since adolescence is a period characterized by significant alterations in sleep/wake patterns and social routines, this period may prove optimal for assessment and treatment of sleep and psychiatric symptoms in those at-risk. The investigators adapted and piloted Interpersonal and Social Rhythm Therapy (IPSRT), an empirically-supported treatment for adults with BP that helps patients stabilize sleep/wake cycles and daily routines, for at-risk adolescents. Preliminary data indicate this approach holds promise for youth at-risk for the development of BP. The investigators also identified intervention for the heterogeneous conditions antecedent to BP as a second path to preventing or delaying BP onset in at-risk youth. The purpose of the proposed study is thus to further develop and examine IPSRT for the adolescent (age 12-18) offspring of parents with BP. The study involves conduct of a small controlled trial (n=50) comparing Brief IPSRT + Data-Informed Referral versus Data-Informed Referral alone to gather preliminary data on feasibility, acceptability and proximal outcomes associated with the intervention. All participants receive a thorough assessment of psychopathology and sleep disturbance (via objective and subjective methods) at baseline, followed by a single feedback session reviewing the findings. As clinically indicated, youth will be offered Data-Informed Referral for any psychiatric symptoms/disorders identified during the intake assessment. Youth will then be randomized to receive either Brief IPSRT or no Brief IPSRT; randomization will be stratified on sleep disturbance and psychopathology. Outcomes will be assessed at 4 time points over 6 months in all participants. Data will be used to inform the design and conduct of a future controlled trial. The proposed approach is in direct accord with strategies outlined in the National Institute of Mental Health (NIMH) Strategic Plan in which the development and testing of innovative interventions to reduce risk and positively alter trajectories of mental illness are informed by research findings regarding robust and malleable risk factors and core features of disease. Research in this area is of great public health importance, as it has the potential to prevent, delay, or ameliorate the progression of this chronic and devastating illness in those at highest risk.

ELIGIBILITY:
Inclusion Criteria:

1. age between 12-18 years;
2. primary residence with a parent or guardian;
3. English language fluency and at minimum a 3rd grade literacy level. Subjects must be able to speak and understand English because one of the study interventions, Brief IPSRT, is an experimental talk-therapy. This therapy cannot practically be translated;
4. a biological parent with a diagnosis of Bipolar Disorder I, II or Not Otherwise Specified (NOS) confirmed via semi-structured diagnostic interview;
5. able and willing to give informed consent/assent to participate.

Exclusion Criteria:

1. a current or lifetime bipolar spectrum disorder diagnosis (i.e., Bipolar Disorder I, II or NOS) by the Schedule for Affective Disorders and Schizophrenia-Present and Lifetime Version (K-SADS-PL);
2. a primary sleep disorder diagnosis by the Structured Interview for DSM-IV Sleep Disorders;
3. current unstabilized psychiatric symptoms as evidenced by a CGI-Severity of > 5 (markedly ill) and/or a C-GAS rating of < 50 (denotes serious symptoms);
4. evidence of mental retardation, pervasive developmental disorder, or organic central nervous system disorder by the K-SADS-PL, parent report, medical history, or school records,
5. a prior course of IPSRT treatment
6. the absence of parental participation for 18 year old potential participants (i.e. 18 year old adolescent subjects need a biological parent with a diagnosis of Bipolar Disorder I, II or Not Otherwise Specified (NOS) to particpate in the study in order for the adolescent to be able to participate) -

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
Change in mood symptom severity | Quarterly over 6 months
  Mood symptom severity assessed via clinical evaluator blind to treatment condition using validated instruments.
Change in sleep | 10 days at intake and 6 months
  actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Tina R Goldstein, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bootzin RR, Stevens SJ. Adolescents, substance abuse, and the treatment of insomnia and daytime sleepiness. Clin Psychol Rev. 2005 Jul;25(5):629-44. doi: 10.1016/j.cpr.2005.04.007. PMID 15953666
- [Background] Frank, E. (2005). Treating bipolar disorder: A clinician's guide to interpersonal and social rhythm therapy. New York: Guilford Press.
- [Background] Frank E, Kupfer DJ, Thase ME, Mallinger AG, Swartz HA, Fagiolini AM, Grochocinski V, Houck P, Scott J, Thompson W, Monk T. Two-year outcomes for interpersonal and social rhythm therapy in individuals with bipolar I disorder. Arch Gen Psychiatry. 2005 Sep;62(9):996-1004. doi: 10.1001/archpsyc.62.9.996. PMID 16143731
- [Background] Goodwin, F. K. & Jamison, K. R. (2007a). Course and outcome. In F.K.Goodwin & K. R. Jamison (Eds.), Manic-depressive illness (2 ed., pp. 119-154). New York: Oxford University Press.
- [Background] Harvey AG. Sleep and circadian rhythms in bipolar disorder: seeking synchrony, harmony, and regulation. Am J Psychiatry. 2008 Jul;165(7):820-9. doi: 10.1176/appi.ajp.2008.08010098. Epub 2008 Jun 2. PMID 18519522
- [Background] Miklowitz DJ, Otto MW, Frank E, Reilly-Harrington NA, Wisniewski SR, Kogan JN, Nierenberg AA, Calabrese JR, Marangell LB, Gyulai L, Araga M, Gonzalez JM, Shirley ER, Thase ME, Sachs GS. Psychosocial treatments for bipolar depression: a 1-year randomized trial from the Systematic Treatment Enhancement Program. Arch Gen Psychiatry. 2007 Apr;64(4):419-26. doi: 10.1001/archpsyc.64.4.419. PMID 17404119
- [Background] Wolfson AR, Carskadon MA. Sleep schedules and daytime functioning in adolescents. Child Dev. 1998 Aug;69(4):875-87. PMID 9768476